CLINICAL TRIAL: NCT02760940
Title: Anemia Treatment in Inflammatory Bowel Disease: Predictive Factors of Response to Oral Iron Treatment
Brief Title: Anemia in Inflammatory Bowel Disease
Acronym: IBD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Juiz de Fora (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAE:0200.0.200.000-10
Record Dates: First submitted 2016-04-27; First posted 2016-05-04 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-05

CONDITIONS: Anemia; Bowel Diseases, Inflammatory
Keywords: Inflammatory bowel diseases; Anemia; Crohn's disease; Ulcerative colitis; Oral iron; Quality of life
MeSH Terms: conditions — Anemia; Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — ferric pyrophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral liposomal iron treatment (Experimental): Oral liposomal iron - 28 mg per day over 8 weeks
  Interventions: Drug: oral liposomal iron

INTERVENTIONS:
Drug: oral liposomal iron — After screening, anemic patients will be treated during 8 weeks with 28mg of oral liposomal iron per day and then the investigators will report data assessing the tolerability and efficacy of oral liposomal iron treatment in these patients.
  Other Names: ferric pyrophosphate

SUMMARY:
Anemia is a clinical manifestation, which is commonly observed in patients with inflammatory bowel disease, and it accounts for significant loss in the quality of life of these patients. The aim of the current study is to assess the effect of orally administered iron treatment, as well as its response predictors in patients with inflammatory bowel disease who are in remission and present anemia. The study will recruit 100 patients with Crohn's disease (CD) and 100 patients with ulcerative colitis (UC) diagnosed and regularly monitored in the Inflammatory Bowel Disease Center at the University Hospital of the Federal University of Juiz de Fora, for clinical, hematological, biochemical and immunological assessment. Blood samples will be collected (10 ml) and the following tests will be performed in all the anemia patients (in remission) at the beginning of the treatment and 8 weeks later: complete blood count, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), erythrocyte sedimentation rate (ESR) , transferrin saturation index, ferritin, serum iron, hepcidin, quantitative C-reactive protein (CRP), interleukin-6 (IL-6)) and fecal calprotectin. In addition, quality of life, anxiety and depression and fatigue questionnaires will be applied to the patients (IBDQ, HAD and Chalder). The World Health Organization (WHO) criteria will be used to diagnose anemia, therefore, hemoglobin lower than 12 g/dl for women and 13g/dl for men will be considered anemia; hemoglobin lower than 10 g/dl will be considered severe anemia. Patients with mild and moderate anemia in remission will be initially treated with oral iron (oral liposomal iron) and the occurrence of possible symptoms related to oral iron intolerance will be assessed, as well as the patients' disease activity level and quality of life. The patients in follow-up will be subjected to new laboratory tests after the eighth oral iron treatment week. The results of the current study are expected to help assessing the oral iron efficacy and response predictors, as well as the side effects of the treatment and its impact on the quality of life of patients.

DETAILED DESCRIPTION:
1. Study Design:

   Two hundred (200) patients with inflammatory bowel disease in remission - 100 patients with Crohn's disease and 100 patients with ulcerative colitis - will be randomly selected.

   The patients will be informed that their participation in the study will generate no expense or financial benefit to them. Any doubts they may have about the study will be clarified and they will be free to participate in it or not. Their refusal will not result in any penalty or change in the way they will be served. They may withdraw their consent or discontinue their participation at any time.

   Laboratory tests will be conducted at the University Hospital, according to the follow-up routine applied to patients with inflammatory bowel disease, and they will represent no risk to health different than that of common blood tests.

   The study protocol will be submitted to the Research Ethics Committee of the University Hospital for evaluation. All patients included in the study will sign a free and informed consent form. The patients will be assessed according to eligibility criteria and their demographic data (age, gender) and body weight will be recorded at the first visit. They will undergo an interview to assess symptoms and possible disease activity one week before the beginning of the treatment. They will also fill out a questionnaire about quality of life, anxiety and depression and another one about fatigue before and after the treatment. Only patients who have completed the 8-week treatment will be included in the study.

   Blood samples (10ml) will be collected for hematological, biochemical and immunological assessments, after the treatment. The following hematological and biochemical tests will be performed in patients with anemia: complete blood count, MCV, MCH, MCHC, ferritin, transferrin saturation index, hepcidin, quantitative CRP, IL-6 and fecal calprotectin.

   The blood collection will be performed by a biochemistry resident at the University Hospital of Juiz de Fora, as well as the examinations, which will be done under the supervision of biochemistry professors of the University Hospital residency program.

   All patients in the study will be subjected to the following tests: a. clinical assessment; b. questionnaire on quality of life c. questionnaire on fatigue d. questionnaire on anxiety and depression e. biochemical assessment; f. ileocolonoscopy with biopsy for histopathological study.
2. Study flowchart

   1. Phase I

      * Patient selection
      * Clinical, biochemical, colonoscopic and histopathological assessment
      * Assessment of IBDQ, HAD and Fatigue scales
   2. Phase II

      * Supplementation with oral iron
      * Monitoring of complications
   3. Phase III

      * Clinical, biochemical, colonoscopic and histopathological reassessment
      * Reassessment of IBDQ, HAD and Fatigue scales
      * Study completion
3. Statistical analysis The collected data will be analyzed by a specific statistical software (SPSS -Statistical Package for Social Sciences™, version 21.0).

The patients will be divided in two groups (mild and moderate anemia) for data analysis, according to their hemoglobin levels. The comparisons between groups, as well as the possible relations between socio-demographic and clinical variables, and changes in IBDQ, HAD and fatigue scales will be analyzed through parametric Student's t-test, Chi-square test or nonparametric Mann-Whitney test, whenever appropriate. Univariate and multivariate logistic analyses will be performed to identify possible independent predictors of oral iron response within the entire group.

The results will be presented as odds ratio (OR) and 95% confidence interval (CI). The statistical significance level will be set at P <0.05, for comparison.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of inflammatory bowel disease (Crohn's disease or ulcerative colitis ) in remission
* Anemia

Exclusion criteria:

* Pre-existing liver disease
* Kidney failure
* Clinically significant pulmonary disease
* Systemic infection
* Pregnancy
* Current history of any type of malignancy (except skin)
* Gastrectomy
* Total colectomy or extensive intestinal resection (> 100 cm )
* Inflammatory bowel disease activity
* Severe anemia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin level improvement | 8 weeks
  The supplementation will be performed in patients with mild to moderate anemia, since patients with severe anemia usually require more aggressive treatments. The replenishment will be provided at no cost to the patients at the dose of 2 (two) iron liposomal iron tablet per day (equivalent to 28 mg of iron). The patients will be instructed to take one tablet of 14 mg twice a day. They will be monitored by telephone in weekly interval periods throughout the intervention phase in order to optimize their adhesion to the treatment and verify the occurrence of possible side effects and the improvement in hemoglobin level.

SECONDARY OUTCOMES:
Improvement of quality of life | 8 weeks
  The IBDQ questionnaire data will be applied before and after treatment. Our study will use the following quality of life classification: Equal to or higher than 200 = Excellent; Between 151 and 199 = Good; Between 101 and 150 = Regular; Lower than or equal to 100 = Poor.
Improvement of fatigue | 8 weeks
  The participants will be instructed to answer the questionnaire on fatigue (Chalder Fatigue Scale - attached) before and 8 weeks after the oral iron treatment.
  The questionnaire comprises 12 items related to the intensity of fatigue symptoms. It is a Likert-type scale with scores ranging from one to four in each item. The items are calculated in bimodal scores. Considering the Likert scale, the values ranging from one to four in bimodal calculations will be considered zero. Values such as three and four will be considered one. The sum in which the value is greater than or equal to four will feature fatigue
Activation of inflammation | 8 weeks
  The inflammatory activity will be assessed according to the Harvey-Bradshaw Index for CD patients and UC patients will be assessed according to the Truelove and Witts criteria.
Improvement of anxiety and depression | 8 weeks
  The participants will be instructed to answer the questionnaire on anxiety and depression (HAD scale) before and 8 weeks after the oral iron treatment.
  The questionnaire comprises 14 items related to anxiety and depression symptoms. It is considered anxiety if obtained 9 or more points, in items of anxiety and no-anxiety if below 8 points. The same criteria is used for depression.

CONTACTS AND LOCATIONS:
Overall Officials: Carla VA Antunes, MSc. MD, Principal Investigator — Federal University of Juiz de Fora

IPD SHARING:
Plan to Share IPD: Yes
data will be published every 6 months until the end of the study

REFERENCES:
- [Background] Bager P, Befrits R, Wikman O, Lindgren S, Moum B, Hjortswang H, Dahlerup JF. The prevalence of anemia and iron deficiency in IBD outpatients in Scandinavia. Scand J Gastroenterol. 2011 Mar;46(3):304-9. doi: 10.3109/00365521.2010.533382. Epub 2010 Nov 15. PMID 21073374
- [Background] Befrits R, Wikman O, Blomquist L, Hjortswang H, Hammarlund P, Bajor A, Klintman D, Blom H. Anemia and iron deficiency in inflammatory bowel disease: an open, prospective, observational study on diagnosis, treatment with ferric carboxymaltose and quality of life. Scand J Gastroenterol. 2013 Sep;48(9):1027-32. doi: 10.3109/00365521.2013.819442. Epub 2013 Jul 29. PMID 23889159
- [Background] Bergamaschi G, Di Sabatino A, Albertini R, Ardizzone S, Biancheri P, Bonetti E, Cassinotti A, Cazzola P, Markopoulos K, Massari A, Rosti V, Porro GB, Corazza GR. Prevalence and pathogenesis of anemia in inflammatory bowel disease. Influence of anti-tumor necrosis factor-alpha treatment. Haematologica. 2010 Feb;95(2):199-205. doi: 10.3324/haematol.2009.009985. Epub 2009 Oct 8. PMID 19815838
- [Background] Gasche C, Ahmad T, Tulassay Z, Baumgart DC, Bokemeyer B, Buning C, Howaldt S, Stallmach A; AEGIS Study Group. Ferric maltol is effective in correcting iron deficiency anemia in patients with inflammatory bowel disease: results from a phase-3 clinical trial program. Inflamm Bowel Dis. 2015 Mar;21(3):579-88. doi: 10.1097/MIB.0000000000000314. PMID 25545376
- [Background] Iqbal T, Stein J, Sharma N, Kulnigg-Dabsch S, Vel S, Gasche C. Clinical significance of C-reactive protein levels in predicting responsiveness to iron therapy in patients with inflammatory bowel disease and iron deficiency anemia. Dig Dis Sci. 2015 May;60(5):1375-81. doi: 10.1007/s10620-014-3460-4. Epub 2014 Dec 12. PMID 25501922
- [Background] Kaitha S, Bashir M, Ali T. Iron deficiency anemia in inflammatory bowel disease. World J Gastrointest Pathophysiol. 2015 Aug 15;6(3):62-72. doi: 10.4291/wjgp.v6.i3.62. PMID 26301120
- [Background] Nemeth E, Rivera S, Gabayan V, Keller C, Taudorf S, Pedersen BK, Ganz T. IL-6 mediates hypoferremia of inflammation by inducing the synthesis of the iron regulatory hormone hepcidin. J Clin Invest. 2004 May;113(9):1271-6. doi: 10.1172/JCI20945. PMID 15124018
- [Background] Nielsen OH, Ainsworth M, Coskun M, Weiss G. Management of Iron-Deficiency Anemia in Inflammatory Bowel Disease: A Systematic Review. Medicine (Baltimore). 2015 Jun;94(23):e963. doi: 10.1097/MD.0000000000000963. PMID 26061331
- [Background] Nielsen OH, Coskun M, Weiss G. Iron replacement therapy: do we need new guidelines? Curr Opin Gastroenterol. 2016 Mar;32(2):128-35. doi: 10.1097/MOG.0000000000000247. PMID 26771951
- [Background] Pisani A, Riccio E, Sabbatini M, Andreucci M, Del Rio A, Visciano B. Effect of oral liposomal iron versus intravenous iron for treatment of iron deficiency anaemia in CKD patients: a randomized trial. Nephrol Dial Transplant. 2015 Apr;30(4):645-52. doi: 10.1093/ndt/gfu357. Epub 2014 Nov 13. PMID 25395392
- [Result] Antunes CV, Hallack Neto AE, Nascimento CR, Chebli LA, Moutinho IL, Pinheiro Bdo V, Reboredo MM, Malaguti C, Castro AC, Chebli JM. Anemia in inflammatory bowel disease outpatients: prevalence, risk factors, and etiology. Biomed Res Int. 2015;2015:728925. doi: 10.1155/2015/728925. Epub 2015 Feb 1. PMID 25705682
- [Result] Filmann N, Rey J, Schneeweiss S, Ardizzone S, Bager P, Bergamaschi G, Koutroubakis I, Lindgren S, Morena Fde L, Moum B, Vavricka SR, Schroder O, Herrmann E, Blumenstein I. Prevalence of anemia in inflammatory bowel diseases in european countries: a systematic review and individual patient data meta-analysis. Inflamm Bowel Dis. 2014 May;20(5):936-45. doi: 10.1097/01.MIB.0000442728.74340.fd. PMID 24572205
- [Result] Bonovas S, Fiorino G, Allocca M, Lytras T, Tsantes A, Peyrin-Biroulet L, Danese S. Intravenous Versus Oral Iron for the Treatment of Anemia in Inflammatory Bowel Disease: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Medicine (Baltimore). 2016 Jan;95(2):e2308. doi: 10.1097/MD.0000000000002308. PMID 26765407